CLINICAL TRIAL: NCT01334112
Title: A Phase II Trial of Axitinib (AG-013736) After Prior Antiangiogenic Therapy in Advanced Hepatocellular Carcinoma
Brief Title: Study of Axitinib in Patients With Unresectable Hepatocellular Carcinoma
Acronym: AXITINIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS515376
Record Dates: First submitted 2011-02-14; First posted 2011-04-12 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Advanced Hepatocellular Carcinoma; Liver Cancer; Axitinib; AG-013736
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib (Experimental): Oral Axitinib (5mg, twice daily) will be administered to all patients
  Interventions: Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Axitinib (AG-013736) — 5mg, oral, twice daily, continuous dosing. A dosing cycle is defined as 4 weeks. Treatment may continue until disease progression/relapse

SUMMARY:
The purpose of this study is to evaluate the potential role of Axitinib (AG-013736) in the treatment of unresectable/metastatic hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
This is a phase II study of an investigational drug, Axitinib following prior antiangiogenic therapy in patients with advanced hepatocellular carcinoma. Hepatocellular carcinoma (HCC) is a primary cancer of the liver. Angiogenesis is a physiological process involving the growth of new blood vessels from pre-existing vessels. A tyrosine kinase is an enzyme that can inhibit angiogenesis. In this study, patients with advanced HCC who have failed prior antiangiogenic therapy, will receive Axitinib in cycles of 4 weeks. Axitinib is an oral, potent and selective inhibitor of angiogenesis. This study will evaluate the response rate of HCC following treatment with Axitinib as well as safety, feasibility, overall survival of patients, progression-free survival, and quality of life in persons with unresectable HCC. The study also compares response determined by RECIST to response determined by Choi Criteria.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable and/or metastatic Hepatocellular Carcinoma
* Previous treatment with tyrosine kinase inhibitors or antiangiogenic drugs
* Life expectancy of ≥12 weeks
* At least one tumor lesion
* At least 2 weeks since the end of prior systemic treatment
* No evidence of pre-existing uncontrolled hypertension
* ECOG 0 or 1
* Adequate organ function
* Not appropriate for curative therapy
* Child A or B7 cirrhosis
* CLIP score ≤ 4

Exclusion Criteria:

* Received any other systemic therapy for Hepatocellular Carcinoma within 2 weeks prior to treatment
* Major surgery <4 weeks or radiation therapy <2 weeks of starting the study treatment
* Previous or concurrent cancer that is distinct in primary site or histology from Hepatocellular Carcinoma
* Severe acute or chronic medical or psychiatric condition
* Need for treatment with prohibited drugs
* Has received local therapy to all measurable lesions
* Stage B8 or higher liver cirrhosis
* Ascites refractory to diuretic therapy
* Clinically significant ECG abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Response rate | Response rate assessed by CT scan at 16 weeks

SECONDARY OUTCOMES:
Feasibility | Assessed at the end of stage 1 (10 patients accrued) and at the end of trial (Stage 2, 29 patients total)
  The ability to administer one or more cycles of Axitinib to >70% of patients at a dose of 5mg po BID
Overall survival | At the completion of trial, 1.5 years
Response rate comparison | Comparison of outcomes with RECIST criteria to Choi criteria and changes to perfusion on DCE ultrasound will occur at the end of stage 1 (after accrual of 10 patients) and trial completion
Progression-free survival | At trial completion, 1.5 years
Quality of life | At completion of trial, 1.5 years
  Assessed by FACT-Hep
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | At completion of trial, 1.5 years
  Efficacy and Toxicity in Asian vs non-Asian patients will be assessed by comparing the adverse effects profile and rate of grade 3 and grade 4 toxicity in these populations
Number of Participants with Adverse Events as a Measure of Safety | At completion of trial, 1.5 years
  Adverse effects profile and rate of grade 3 and 4 toxicity will be assessed as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MSc, FRCPC, MD, Principal Investigator — University Health Network, Princess Margaret Hospital; Kelly Burak, MD, FRCPC, BSc, MSc, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Hospital, Alberta Health Services, Calgary, Alberta
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario